CLINICAL TRIAL: NCT03553056
Title: Feasibility of a Smart-phone Based Support System for Hazardous Drinkers
Acronym: NZStepAway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Waitemata District Health Board (Other Government); University of Alaska Anchorage (Other)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: U1111-1195-2467
Record Dates: First submitted 2018-05-20; First posted 2018-06-12 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Consumption
Keywords: alcohol; hazardous drinking; mobile phone app; clinical trial
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): NZ Step Away app
  Interventions: Other: NZ Step Away app
- Control (Active Comparator): Modified NZ Step Away app
  Interventions: Other: Modified NZ Step Away app

INTERVENTIONS:
Other: NZ Step Away app — Access to 10 modules of the app (namely: drinkers profile, goal setting, rewards, cravings, strategies, support, reminders, high risk times, moods, activities)
  Arms: Intervention
Other: Modified NZ Step Away app — Access to 2 modules of the app (namely: drinkers profile and goals setting)
  Arms: Control

SUMMARY:
A feasibility trial to determine whether six months access to the New Zealand 'Step Away' app can reduce the frequency of alcohol abuse and increase engagement with substance abuse-related health services by hazardous drinkers

DETAILED DESCRIPTION:
Rationale: Hazardous drinking is an established drinking pattern that carries a risk of harming the drinker's physical and psychological health, and/or having a harmful social effect on the drinker, their families and the community. Interventions to support people who are drinking at hazardous levels are proven to be beneficial and cost-effective at both individual and population levels. However, very few people report having received help to reduce their alcohol consumption, despite support being available. Those who do seek help predominantly talk to their GP first, who then refers them for specialist support. Consequently, there remains a significant gap between the population 'in need' of treatment and those actually engaged in treatment. Mobile-phone based alcohol interventions have the potential to function as a stand-alone intervention to help people address their alcohol problem, and/or act as a conduit to more intensive treatment. 'Step Away' is a smartphone-delivered health intervention designed in the USA to help individuals moderate or abstain completely from drinking alcohol. It is the only alcohol-related mobile app whose development was informed by an empirically-supported intervention grounded in a psychological theory. While the app has shown promise in a North American sample, a well-powered clinical trial of the intervention has yet to be undertaken. In its current form the app is not suitable for adoption in New Zealand as it uses North American drinking norms and safe drinking guidelines, numerous "Americanisms" and the imperial measurement system, and it focuses on US care services. However, a New Zealand version of 'Step Away' could easily be developed, with input from New Zealand stakeholders and end-users.

Aims: To 1) adapt the "Step Away' app for New Zealand, then 2) undertake a feasibility study to determine whether six months access to the app can reduce the frequency of alcohol abuse and increase engagement with substance abuse-related health services in adult, hazardous drinkers in Auckland.

Design: Double-blind, randomised-controlled trial.

Recruitment: Community advertising, including social media.

Sample size: As a feasibility study, no sample size calculation was undertaken. However, 200 people (100 in each arm) will provide sufficient data to ascertain the direction and likely effect size for the various alcohol-related outcomes, the likely recruitment rate, and estimates around participant retention.

ELIGIBILITY:
Inclusion Criteria:

* reside in Auckland, New Zealand
* at least 18 years of age
* have access to a smartphone
* report that they currently drink alcohol
* have had at least two episodes of binge drinking (defined as six or more drinks on one occasion) in the past 30 days
* meet the criteria for hazardous drinking (i.e. 8-19 on the AUDIT)
* express motivation to moderate or abstain from drinking.

Exclusion Criteria:

* Identified during screening as having moderate to severe alcohol dependence (≥20 score on the AUDIT)
* Currently enrolled in an alcohol programme
* Another person in the household is already a participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Number of days spent hazardously drinking in the last 30 days | Measured at 6 months post-randomization

SECONDARY OUTCOMES:
Number of days spent hazardously drinking in the last 30 days | Measured at 3 months post-randomization
Number of days spent hazardously drinking in the last 30 days | Measured at 1 month post-randomization
Percentage of days spent hazardously drinking in the last 30 days | Measured at 6 months post-randomization
Percentage of days spent hazardously drinking in the last 30 days | Measured at 3 months post-randomization
Percentage of days spent hazardously drinking in the last 30 days | Measured at 1 month post-randomization
Drinks per day over the last 30 days | Measured at 6 months post-randomization
Drinks per day over the last 30 days | Measured at 3 months post-randomization
Drinks per day over the last 30 days | Measured at 1 month post-randomization
Drinking-related problems | Measured at 6 months post-randomization
  Measured by the Short Inventory of Problems - Revised (SIP-R)
Any contact with substance abuse-related health services since randomization | Measured at 6 months post-randomization
  Measured as 'Yes' or 'No'
Any contact with substance abuse-related health services since randomizations | Measured at 3 month post-randomization
  Measured as 'Yes' or 'No'
Any contact with substance abuse-related health services since randomization | Measured at 1 month post-randomization
  Measured as 'Yes' or 'No'
Any contact with substance abuse-related health services since randomization | Measured at 2 weeks post-randomization
  Measured as 'Yes' or 'No'
Who they have talked to about their drinking, since randomization | Measured at 6 months post-randomization
  'Yes' or 'No' answers to options of 'Partner, Family, Whanau, GP/Doctor, Other'
Who they have talked to about their drinking, since randomization | Measured at 3 months post-randomization
  'Yes' or 'No' answers to options of 'Partner, Family, Whanau, GP/Doctor, Other'
Who they have talked to about their drinking, since randomization | Measured at 1 month post-randomization
  'Yes' or 'No' answers to options of 'Partner, Family, Whanau, GP/Doctor, Other'
Who they have talked to about their drinking, since randomization | Measured at 2 weeks post-randomization
  'Yes' or 'No' answers to options of 'Partner, Family, Whanau, GP/Doctor, Other'
Serious adverse events | Measured at 6 months post-randomization
Serious adverse events | Measured at 3 months post-randomization
Serious adverse events | Measured at 1 month post-randomization
Serious adverse events | Measured at 2 weeks post-randomization
App utlization | Measured at 6 months post-randomization
App utlization | Measured at 3 months post-randomization
App utlization | Measured at 1 month post-randomization
App utlization | Measured at 2 weeks post-randomization
Withdrawal from study | Measured at 6 months post-randomization
Withdrawal from study | Measured at 3 months post-randomization
Withdrawal from study | Measured at 1 month post-randomization
Withdrawal from study | Measured at 2 weeks post-randomization
Loss to follow-up | Measured at 6 months post-randomization
Loss to follow-up | Measured at 3 months post-randomization
Loss to follow-up | Measured at 1 month post-randomization
Loss to follow-up | Measured at 2 weeks post-randomization
Alcohol withdrawal | Measured at 6 months post-randomization
  Experience of any specific signs and symptoms (i.e. shakiness, sweating, vomiting, fast heart rate, mild fever, seizures, seeing or hearing things that others do not, confusion, shivering, other) since randomization, that may be due to changing the amount of alcohol consumed. Recorded as: not at all, mild, moderate, severe.
Alcohol withdrawal | Measured at 3 months post-randomization
  Experience of any specific signs and symptoms (i.e. shakiness, sweating, vomiting, fast heart rate, mild fever, seizures, seeing or hearing things that others do not, confusion, shivering, other) since randomization, that may be due to changing the amount of alcohol consumed. Recorded as: not at all, mild, moderate, severe.
Alcohol withdrawal | Measured at 1 month post-randomization
  Experience of any specific signs and symptoms (i.e. shakiness, sweating, vomiting, fast heart rate, mild fever, seizures, seeing or hearing things that others do not, confusion, shivering, other) since randomization, that may be due to changing the amount of alcohol consumed. Recorded as: not at all, mild, moderate, severe.
Alcohol withdrawal | Measured at 2 weeks post-randomization
  Experience of any specific signs and symptoms (i.e. shakiness, sweating, vomiting, fast heart rate, mild fever, seizures, seeing or hearing things that others do not, confusion, shivering, other) since randomization, that may be due to changing the amount of alcohol consumed. Recorded as: not at all, mild, moderate, severe.
Medical help sought for any moderate-severe alcohol withdrawal signs and symptoms | Measured at 6 months post-randomization
  Measured as 'Yes' or 'No'
Medical help sought for any moderate-severe alcohol withdrawal signs and symptoms | Measured at 3 months post-randomization
  Measured as 'Yes' or 'No'
Medical help sought for any moderate-severe alcohol withdrawal signs and symptoms | Measured at 1 month post-randomization
  Measured as 'Yes' or 'No'
Medical help sought for any moderate-severe alcohol withdrawal signs and symptoms | Measured at 2 weeks post-randomization
  Measured as 'Yes' or 'No'
Still experiencing any moderate-severe alcohol withdrawal signs and symptoms | Measured at 6 months post-randomization
  Measured as 'Yes' or 'No'
Still experiencing any moderate-severe alcohol withdrawal signs and symptoms | Measured at 3 months post-randomization
  Measured as 'Yes' or 'No'
Still experiencing any moderate-severe alcohol withdrawal signs and symptoms | Measured at 1 month post-randomization
  Measured as 'Yes' or 'No'
Still experiencing any moderate-severe alcohol withdrawal signs and symptoms | Measured at 2 weeks post-randomization
  Measured as 'Yes' or 'No'

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- National Institute for Health Innovation, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No